CLINICAL TRIAL: NCT00105833
Title: Improving Outcomes of Depression in Primary Care
Acronym: DEP-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHI 20-020
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2009-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Multifaceted collaborative intervention for depression based in primary care
  Interventions: Behavioral: Collaborative Care - Depression Decision Support (DDS)
- Arm 2 (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Collaborative Care - Depression Decision Support (DDS) — Multifaceted collaborative intervention for depression based in primary care
  Other Names: Depression Decision Support (DDS)
  Arms: Arm 1

SUMMARY:
Depression is common in primary care settings, and associated with substantial physical and psychosocial impairment and increased healthcare utilization. Despite efforts to educate primary care providers, depression is often undetected or undertreated in primary care settings. The main objective of this study was to determine the impact of a low-intensity, care management intervention on depression treatment outcomes of patients in a VA primary care setting.

DETAILED DESCRIPTION:
OBJECTIVE(S): The primary objective of the study was to determine the impact of a low-intensity, care management intervention on depression treatment outcomes of patients in a VA primary care setting. Secondary objectives were to determine the extent to which primary care clinicians adhere to major depression treatment guidelines, the extent to which the intervention impacts healthcare utilization, and to examine the impact of provider and patient covariates (including pain and adherence) on depression treatment response PLAN: Randomized controlled trial. METHODS: All clinicians first participated in the MacArthur Depression Education Program (DEP). After stratification by discipline and site, clinicians were randomized to receive the Depression Decision Support (DDS) intervention versus usual care (which included an on-site mental health team). Patients were nested within clinician intervention status. DDS intervention clinicians received serial reports of depression severity scores and other clinical data for their enrolled patients. The DDS care manager made one telephone contact with each intervention patient, and invited patients to attend a depression group education session. The DDS team monitored patient depression severity over time, and targeted additional time and effort towards patients not showing improvement. Additional DDS intervention included making further recommendations to primary care clinicians, and in some cases, a one-time consultation with the DDS psychiatrist.

Potential subjects were identified from lists of patients due for appointments with primary care clinicians, and were contacted for telephone screening. Patients were enrolled if they had Patient Health Questionnaire (PHQ-9) scores >10 or a Hopkins Symptom Checklist (SCL-20) score of > 1.0 at a subsequent in-person interview. There were no restrictions by age or sex. Patients were excluded if they had psychotic symptoms, dementia, serious suicidal ideation, very severe depression (PHQ-9 >25), or had been treated by mental health clinicians within the previous six months. The intervention lasted 12 months. Depression symptom severity (SCL-20) and health related quality of life (SF-36V) at 6 and 12-months were primary outcomes. Primary analyses employed mixed-model repeated measure analyses of covariance, which include a random effect for clinician and fixed effects for time and intervention status.

FINDINGS TO DATE: Five Portland VA clinic sites and 41 clinicians participated. 3,103 patients were screened, and 402 patients were enrolled. Three hundred seventy-five met final eligibility criteria. There were no adverse events. SCL-20 scores improved in both groups over 12 months (slope: -.382; 95% CI -.488, -.276), but there was no effect of the intervention on SCL-20 or Short Form-36V compared to usual care. There was greater initial improvement in PHQ-9 for intervention patients (p=.030); however, this effect diminished over time. At 12 months, intervention patients reported greater satisfaction (p=.002), and were more likely to have received antidepressants. To date, 10 manuscripts supported by the project have been published. One manuscript examining associations between stressful live events and depression outcomes has been submitted for publication.

ELIGIBILITY:
Inclusion Criteria:

Primary care patients of eligible providers with depression (Patient Health Questionnaire [PHQ-9] depression scores of 10 to 25 or Hopkins Symptom Checklist-20 [SCL-20] scores >= 1.0)

Exclusion Criteria:

Patients who had received treatment from mental health specialists within the previous 6 months; who had received a diagnosis of psychotic disorder, dementia, or bipolar disorder; or who were considered to be terminally ill

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2002-07; Primary Completion 2004-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Symptom Checklist SCL-20 score | SCL-20 score over 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Dobscha, MD, Principal Investigator — VA Portland Health Care System, Portland, OR; Martha S. Gerrity, MD MPH PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

REFERENCES:
- [Result] Snyder K, Dobscha SK, Ganzini L, Hoffman WF, Delorit MA. Clinical outcomes of integrated psychiatric and general medical care. Community Ment Health J. 2008 Jun;44(3):147-54. doi: 10.1007/s10597-007-9117-4. Epub 2007 Dec 11. PMID 18071900
- [Result] Williams JW Jr, Gerrity M, Holsinger T, Dobscha S, Gaynes B, Dietrich A. Systematic review of multifaceted interventions to improve depression care. Gen Hosp Psychiatry. 2007 Mar-Apr;29(2):91-116. doi: 10.1016/j.genhosppsych.2006.12.003. PMID 17336659
- [Result] Dobscha SK, Corson K, Pruitt S, Crutchfield M, Gerrity MS. Measuring depression and pain with home health monitors. Telemed J E Health. 2006 Dec;12(6):702-6. doi: 10.1089/tmj.2006.12.702. PMID 17250493
- [Result] Dobscha SK, Corson K, Hickam DH, Perrin NA, Kraemer DF, Gerrity MS. Depression decision support in primary care: a cluster randomized trial. Ann Intern Med. 2006 Oct 3;145(7):477-87. doi: 10.7326/0003-4819-145-7-200610030-00005. PMID 17015865
- [Result] Gerrity MS, Corson K, Dobscha SK. Screening for posttraumatic stress disorder in VA primary care patients with depression symptoms. J Gen Intern Med. 2007 Sep;22(9):1321-4. doi: 10.1007/s11606-007-0290-5. Epub 2007 Jul 17. PMID 17634781
- [Result] Dobscha SK, Corson K, Gerrity MS. Depression treatment preferences of VA primary care patients. Psychosomatics. 2007 Nov-Dec;48(6):482-8. doi: 10.1176/appi.psy.48.6.482. PMID 18071094
- [Result] Dobscha SK, Winterbottom LM, Snodgrass LS. Reducing drug costs at a Veterans Affairs hospital by increasing market-share of generic fluoxetine. Community Ment Health J. 2007 Feb;43(1):75-84. doi: 10.1007/s10597-006-9062-7. Epub 2006 Sep 22. PMID 17029000
- [Result] Corson K, Gerrity MS, Dobscha SK. Screening for depression and suicidality in a VA primary care setting: 2 items are better than 1 item. Am J Manag Care. 2004 Nov;10(11 Pt 2):839-45. PMID 15609737
- [Result] Dobscha SK, Corson K, Solodky J, Gerrity MS. Use of videoconferencing for depression research: enrollment, retention, and patient satisfaction. Telemed J E Health. 2005 Feb;11(1):84-9. doi: 10.1089/tmj.2005.11.84. PMID 15785225
- [Result] Dobscha SK, Anderson TA, Hoffman WF, Winterbottom LM, Turner EH, Snodgrass LS, Hauser P. Strategies to decrease costs of prescribing selective serotonin reuptake inhibitors at a VA Medical Center. Psychiatr Serv. 2003 Feb;54(2):195-200. doi: 10.1176/appi.ps.54.2.195. PMID 12556600
- [Result] Dobscha SK, Gerrity MS, Corson K, Bahr A, Cuilwik NM. Measuring adherence to depression treatment guidelines in a VA primary care clinic. Gen Hosp Psychiatry. 2003 Jul-Aug;25(4):230-7. doi: 10.1016/s0163-8343(03)00020-3. PMID 12850654